CLINICAL TRIAL: NCT07174258
Title: The Effect of Different Myofascial Release Techniques on Flexibility, Balance, and Performance In Individuals With Hamstring Shortness
Brief Title: Myofascial Release Wıth Hamstring Shortness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ayca Nur Kilinc, Msc, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3737
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Myofacial Pain
Keywords: balance; manual myofascial relasing; performance
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): (Manual Myofascial Relasing group
  Interventions: Other: Manual myofascial release group
- Group II (Experimental): Graston Group
  Interventions: Other: Graston group
- Group III (Experimental): Home based exercise group
  Interventions: Other: Home based exercise group

INTERVENTIONS:
Other: Manual myofascial release group — Manual myofascial release techniques were applied to Group I on the feet, legs, and thighs, twice a week for 4 weeks.
  Arms: Group I
Other: Graston group — Graston was applied to the gastrocnemius and hamstring muscles, and before the application, solid petroleum jelly was applied to the area to lubricate the surface. A stainless steel Graston instrument was used for the application, using a superficial sweep technique at a 30-degree angle for 2 minutes, followed by a deep sweep for 30 seconds.
  Arms: Group II
Other: Home based exercise group — Group III received a home exercise program that included stretching exercises. They were asked to perform the exercises twice a week for four weeks, with 15-20 repetitions, without any intervention from a physiotherapist.
  Arms: Group III

SUMMARY:
The aim of this study will be to investigate the effects of different myofascial release techniques on flexibility, balance, and performance in individuals with hamstring (HT) muscle shortness. A total of 48 participants with hamstring shortness will be randomly assigned into three groups: Group I (Manual Myofascial Release Group), Group II (Graston Group), and Group III (Home Exercise Group).

DETAILED DESCRIPTION:
The aim of this study will be to investigate the effects of different myofascial release techniques on flexibility, balance, and performance in individuals with hamstring (HT) muscle shortness. A total of 48 participants with hamstring shortness will be randomly assigned into three groups: Group I (Manual Myofascial Release Group), Group II (Graston Group), and Group III (Home Exercise Group). The Graston and manual myofascial release groups will receive interventions twice a week for 4 weeks, totaling 8 sessions, in addition to being provided with a home exercise brochure. The home exercise group will receive only the brochure. All participants will be evaluated in terms of balance, flexibility, and performance both before and after the interventions. Balance will be assessed using the Single Leg Stance Test (SLST) and the Y Balance Test (YBT); flexibility will be assessed using the V Sit and Reach Test; agility and performance will be assessed using the Illinois Agility Test and the T-Drill Test.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 60 years of age,
* Visible shortening of the hamstring muscle,
* Passive straight leg raise (SLR) angle ≤ 70 degrees,
* No musculoskeletal problems in the lower extremity,
* First-time applicant for treatment of hamstring tightness, and
* Volunteering to participate in the study

Exclusion Criteria:

* Participating in intense physical activity within the last 24 hours
* Having had previous lower extremity trauma or surgery
* Having ankle instability
* Having neurological findings during the DBK test
* Having used analgesic, anti-inflammatory, or muscle relaxant medications within the last month
* Having obesity, diabetes, and/or metabolic syndrome
* Being pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
V-Sit-Reach Test | at the beginning of the study and 4 weeks after the start
  This test can be easily performed without requiring a flexibility bench. The subject is asked to sit with their heels touching the floor and their toes pointing upward, with a distance of 30 cm between their feet. A straight line is drawn between their heels, which is considered the zero point. The subject reaches forward toward their heels without bending their knees. The best measurement is recorded as + or -.
Single Leg Stance Test | at the beginning of the study and 4 weeks after the start
  It's one of the most frequently used tests by physiotherapists to assess postural stability. During the test, the patient is asked to keep their eyes open and their hands secured at the waist. They are asked to stand on one leg without any support, with the raised leg not touching the ground and avoiding any jumping, hopping, or other similar movements. This test is performed three times on each leg, and the average is calculated.
Y Balance Test | at the beginning of the study and 4 weeks after the start
  The Y-shaped dynamic balance test is both economical and easy to perform compared to other balance tests and is an effective test for determining balance asymmetry. The Y-shaped balance test assesses individuals' dynamic balance in the anterior, posteromedial, and posterolateral directions. Before starting the test, the Y-shaped directions are determined. The average of the three distances is taken, and the ratio of the absolute distance to leg length is recorded.
T Drill Test | at the beginning of the study and 4 weeks after the start
  Four cones are required for the course. Participants begin at cone "A" at the start command. They run straight to cone "B" and touch it with their right hand. They then sidestep to cone "C" and touch it with their left hand. They then sidestep to cone "D" and touch it with their right hand. Finally, they sidestep to cone "B" and touch it with their left hand. They then run back to cone "A" and stop the stopwatch as soon as they reach cone "A." The time is recorded in seconds. They run three times, resting between each repetition, and their best time is recorded.
Illinois Agility Test | at the beginning of the study and 4 weeks after the start
  The Illinois test is administered to measure agility levels by considering individuals' ability to change direction. Before the test, participants are provided with the necessary information, and the course is explained in detail. Before starting the test, participants are given the opportunity to complete 3-4 trials at a slow pace. The test course is 5 meters wide and 10 meters long, with cones arranged 3.3 meters apart in the center.
  This test consists of a 40-meter straight run and a 20-meter slalom run between cones, with 180-degree turns every 10 meters. After a full rest, the test is administered twice, and the best result is recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yılmaz Menek, PhD, Study Director — Medipol University